CLINICAL TRIAL: NCT02196844
Title: Couple-Based Yoga Program for Patients Receiving Thoracic Radiation and Their Family Caregivers
Brief Title: Yoga Program for Lung Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-0036; 1K01AT007559-01A1 (NIH); NCI-2015-01902 (Other: NCI CTRP)
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Hatha Yoga; Questionnaires; Surveys; Walk Test; Caregiver
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga Group (Experimental): Couple-Based Hatha Yoga Program: 5-6 weeks of a yoga program, three sessions per week (up to 15 sessions) during radiation treatment. At fifth session, CD given for practicing yoga at home. 10 questionnaires completed before first radiation treatment, each week during radiation, 5 questionnaires halfway through radiation treatment schedule. at radiation treatment completion, and again 3 months later. Saliva samples to measure the level of cortisol collected at baseline visit, at end of treatment, and 3 months after radiation therapy. 6-minute walk test performed at baseline, at the end of radiation therapy, and 3 months after radiation therapy.
  Interventions: Behavioral: Hatha Yoga; Behavioral: Questionnaires; Other: Walk Test
- Wait-List Control Group (Experimental): 10 questionnaires completed before first radiation treatment, each week during radiation, 5 questionnaires halfway through radiation treatment schedule, at radiation treatment completion, and again 3 months later. Saliva samples to measure the level of cortisol collected at baseline visit, at end of treatment, and 3 months after radiation therapy. 6-minute walk test performed at baseline, at the end of radiation therapy, and 3 months after radiation therapy.
  Participants given the option to take part in the couple-based Hatha Yoga program (off study) after they finish their last questionnaire packet.
  Interventions: Behavioral: Questionnaires; Other: Walk Test
- Caregivers (Experimental): Yoga Group - Caregivers: 5-6 weeks of yoga during patient's radiation treatment. At fifth session, caregiver given CD for practicing yoga at home. During each week of patient's radiation, caregiver completes questionnaire about their feelings about yoga sessions. 10 questionnaires completed before patient's first radiation treatment, each week during radiation, 5 halfway through radiation, at radiation completion, and again 3 months later. Saliva samples collected at baseline visit, at end of treatment, and 3 months after patient's radiation therapy.
  Waitlist-Control Group - Caregivers: 10 questionnaires completed before patient's first radiation treatment, each week during radiation, 5 halfway through radiation. at radiation completion, and again 3 months later. Saliva samples collected at baseline visit, at end of treatment, and 3 months after radiation therapy.
  Caregivers given option to take part in yoga program after they finish their last questionnaire packet.
  Interventions: Behavioral: Hatha Yoga; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Hatha Yoga — 5-6 weeks of a couple-based yoga program, three sessions per week (up to 15 sessions) during radiation treatment.
  Arms: Caregivers; Yoga Group
Behavioral: Questionnaires — 10 questionnaires completed before first radiation treatment, each week during radiation, 5 questionnaires halfway through radiation treatment schedule. at radiation treatment completion, and again 3 months later.
  Other Names: Surveys
Other: Walk Test — 6-minute walk test performed at baseline, at the end of radiation therapy, and 3 months after radiation therapy.
  Arms: Wait-List Control Group; Yoga Group

SUMMARY:
The goal of this behavioral research study is to learn the opinion of patients and their caregivers about a couple-based Hatha Yoga program (Group 1) during treatment for cancer. Researchers also want to learn the effect of this program on lung function, distress, biological function, and quality of life. For comparison purposes, there will also be a group of participants (Group 2) that does not take part in this program.

You and your caregiver/family member will have about a 50/50 chance of being assigned to each group. The groups are randomly assigned, but it is also based on other factors such as your age and the status of the disease.

DETAILED DESCRIPTION:
Caregiver:

If you agree to take part in this study, your demographic information (such as your age, sex, and race) will be recorded. You will then be assigned to 1 of 2 study groups:

* If you are in Group 1, you will take part in the couple-based Hatha Yoga program.
* If you are in Group 2, you will not take part in the couple-based Hatha Yoga program but will complete the same study procedures as Group 1. You will be given the option to take part in the couple-based Hatha Yoga program (off study) after you finish your last questionnaire packet.

You and the patient will have about a 1 in 2 chance of being assigned to each group (as in the flip of a coin). The groups are randomly assigned, but the assignment will also depend on the age, sex, and status of disease of the patient.

Yoga Sessions:

If you are in Group 1, you will take part in up to 15 sessions of Hatha yoga with the patient over the course of radiation therapy (2-3 weekly sessions). Each 45- to 60-minute session will be guided by an instructor. You should attend each session with the patient.

During the yoga sessions, you will be asked to do deep-breathing exercises and perform different stretching and movement exercises. The movements are designed not to be difficult, and you will sit on the floor or in a chair while you do them. You can move through the exercises at your own pace. The instructor will be available to answer any question you may have about the practice of Hatha yoga. Most of the yoga sessions may be videotaped. This is so the researchers can keep track of the quality of the sessions. Only the study staff will be able to view this videotape. The video files are digital and will be deleted after all the data are studied.

At your fifth session, you will be given a CD and instructions for practicing Hatha yoga at home. While the patient is receiving radiation therapy, you will be asked to practice at home 1 time a day either with him/her or alone on the days you do not have a session at the clinic. Your answers to the questions will not be shared with the patient.

During each week of radiation therapy, you will also complete a questionnaire about your feelings about the Hatha Yoga sessions. You will be asked to list what you liked or disliked, what you found most and least useful, and how you would rate the instructor. You will also be asked about how often you practice outside of class and if you think you are benefitting from the Hatha Yoga program. It should take about 5 minutes to complete this questionnaire.

Questionnaires for All Study Participants:

You will complete about 10 questionnaires before the patient's first radiation treatment, at the end of the treatment (usually 6 weeks later), and then again 3 months later. The questionnaires have questions about your mood, your quality of life, your feelings about being a caregiver, and your relationship with the patient. It should take about 45 minutes to complete these questionnaires each time.

You will also complete about 5 questionnaires halfway through the radiation treatment schedule. These questionnaires have questions about your quality of life. These should take about 20 minutes to complete.

Saliva Testing for All Study Participants:

After your first visit, at the end of the patient's radiotherapy, and 3 months after the radiation, you will be asked to provide saliva samples to measure the level of cortisol (a stress hormone). These saliva samples will be collected 4 times a day for 2 days in a row. You will be asked to collect the samples when you first wake up, about 45 minutes later, about 10 hours after waking, and then at bedtime. To collect each saliva sample, you will chew on a cotton ball for a few seconds and then put the cotton in a small plastic tube. You will write down the times at which you took these samples. You will then either bring the samples into the clinic or mail the samples back to MD Anderson in postage-paid envelopes that will be provided to you. The supplies needed for this testing will also be provided at no cost to you. These saliva samples will be destroyed after being studied.

Follow-Up Phone Calls:

If you are in Group 1, after you have completed the weekly yoga classes, you will receive phone calls from a study team member asking about your at home Hatha Yoga practice. You will be called every other week between the end of your radiotherapy and your final visit with the study. This will be about 5-6 phone calls and they will last approximately 10 minutes each.

Length of Study:

Your participation on this study will be over when you have completed the questionnaires at the time of the patient's 3-month follow-up appointment in the thoracic clinic.

This is an investigational study.

Up to 50 patients and their family members, for a total of 100 participants, will take part in this study. All will be enrolled at MD Anderson.

Patients:

If you agree to take part, your medical history and demographic information (such as your age, sex, and race) will be recorded. By signing this consent, you also agree that your caregiver will be approached to take part in this study.

After your first visit, you will be randomly assigned (as in the roll of dice) to 1 of 2 groups:

* Group 1 will take part in the couple-based Hatha Yoga program.
* Group 2 will not take part in the couple-based Hatha Yoga program but will complete the same procedures as group 1. Participants in this group will be given the option to take part in the couple-based Hatha Yoga program (off study) after they finish their last questionnaire packet.

Group 1:

Hatha Yoga Sessions:

You and your caregiver have a 50/50 chance to be assigned to the intervention group or to the usual care group. If you are assigned to the intervention group, you will take part in up to 15 sessions of Hatha yoga over the course of radiation therapy (2-3 weekly sessions). Each 45- to 60-minute session will be guided by an instructor. You should attend each session together as a couple.

During the yoga sessions, you will be asked to do deep-breathing exercises and perform different stretching and movement exercises. The movements are designed not to be difficult, and you will sit on the floor or in a chair while you do them. You can move through the exercises at your own pace. The instructor will be available to answer any questions you may have about the practice of Hatha yoga. Most of the yoga sessions may be videotaped. This is so the researchers can keep track of the quality of the sessions. Only the study staff will be able to view this videotape. The video files are digital and will be deleted after all the data are studied.

At your fifth session, you will be given a CD and instructions for practicing Hatha yoga at home. While you are receiving radiation therapy, you will be asked to practice at home 1 time a day either with your caregiver or alone on the days you do not have a session at the clinic.

If you are assigned to the yoga group, during each week of radiation therapy, you will also complete a questionnaire asking your feelings about the Hatha Yoga sessions. You will be asked to list what you liked or disliked, what you found most and least useful, and how you would rate the instructor. You will also be asked about how often you practice outside of class and if you think you are benefitting from the Hatha Yoga program. It should take about 5 minutes to answer this questionnaire. Your answers to the questions will not be shared with your caregiver.

Groups 1 and 2:

Questionnaires:

You will complete about 10 questionnaires before your first radiation treatment and again after you complete your treatment schedule (usually 6 weeks later) and then again 3 months later. The questionnaires ask about your health, any symptoms you may be having, your mood, your level of fatigue, your sleeping habits, your relationship, and your quality of life. It should take about 45 minutes to complete these questionnaires.

You will also complete about 5 questionnaires again halfway through your radiation treatment schedule. These questionnaires ask about your quality of life. These should take about 20 minutes to complete.

Follow-Up Phone Calls:

If you are in Group 1, after you have completed the weekly yoga classes, you will receive phone calls from a study team member asking about your at home Hatha Yoga practice. You will be called every other week between the end of your radiotherapy and your final visit with the study. This will be about 5-6 phone calls and they will last approximately 10 minutes each.

Saliva Testing:

After your baseline visit, at the end of treatment, and 3 months after radiotherapy, you will be asked to provide saliva samples to measure the level of cortisol (a stress hormone). These saliva samples will be collected 4 times a day for 2 days in a row. You will be asked to collect the samples when you first wake up, about 45 minutes later, about 10 hours after waking, and then at bedtime. To collect each saliva sample, you will chew on a cotton ball for a few seconds and then put the cotton in a small plastic tube. You will write down the times at which you took these samples. You will then either either bring the samples into the clinic or mail the samples back to MD Anderson in postage-paid envelopes that will be provided to you. The tubes will also be provided at no cost to you. These saliva samples will be sent to These saliva samples will be destroyed after being studied.

Lung Function tests:

Pulmonary Function tests (PFTs) are part of your standard treatment as a patient at MD Anderson. We will request copies of these, as available, from your electronic medical records at baseline and 3 months after radiotherapy.

You will also complete the 6-minute walking test. The six-minute walk test measures the distance you are able to walk over a total of six minutes on a hard, flat surface. The goal is to walk as far as possible in six minutes. You will be allowed to self-pace and rest as needed during the walk along a marked walkway. You will complete a 6-minute walk at baseline, at the end of radiotherapy, and 3 months after radiotherapy.

Length of Study:

Your participation on this study will be over when you have completed the questionnaires at the time of your 3-month follow-up appointment in the thoracic clinic.

This is an investigational study.

Up to 50 patients and their caregivers, for a total of 100 participants, will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lung or esophageal cancer stages I through IIIB who are going to receive at least 5 weeks of daily thoracic radiation therapy with or without chemotherapy in the Department of Radiation Oncology at M. D. Anderson Cancer Center (MDACC) and have an eligible and consenting family caregiver living with the patient while he/she receives treatment (i.e., adult child, sibling, parent).
2. Patients and caregivers must both be at least 18 years old and able to give informed consent.
3. Patients and caregivers must be able to read, write, and speak English.
4. Patient and caregiver must be willing to be videotaped.

Exclusion Criteria:

1. Patients and caregivers who are not oriented to time, place, and person.
2. Patients who have regularly practiced yoga in the year prior to recruitment.
3. Patients who have an ECOG performance status score greater than 2 at time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of Couple-Based Yoga (VKC) in Lung Cancer Patients and Caregivers | 6 weeks
  Feasibility determined by 3 criteria:
  1) accrual of sample within 2 years; 2) adherence, retention and satisfaction rates; and 3) no serious adverse events that are directly attributable to the intervention. Trial judged feasible if at least: 50% of eligible dyads agree to randomization and enroll, 70% of enrolled dyads complete the study and at least 10 yoga sessions have been attended, and 75% of participants rate the program as "useful" or "very useful". Study conditions recruitment rate, drop-out rates, and completion rates calculated along with 95% confidence intervals (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, PHD, MA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org